CLINICAL TRIAL: NCT04761380
Title: Decreased Tongue Strength is Related to Skeletal Muscle Mass in COPD Subjects
Status: Completed | Type: Observational
Sponsor: Kindai University (Other)
Responsible Party: Sponsor
Other Study IDs: 0414
Record Dates: First submitted 2020-10-09; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dysphagia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stable COPD subjects
  Interventions: Diagnostic Test: balloon-based tongue pressure measurement device
- age-matched control subjects subjects who did not have any pulmonary disease
  Interventions: Diagnostic Test: balloon-based tongue pressure measurement device

INTERVENTIONS:
Diagnostic Test: balloon-based tongue pressure measurement device — The probe was inflated at a baseline pressure of 19.6 kilopascal (kPa). To measure MTP, the balloon was positioned on the anterior palate with the lips closed. Subjects raised their tongue and compressed the balloon onto the palate with maximal voluntary muscular effort for approximately 7s. The measurement was taken three times with a 1-min interval. The maximum value was recorded as the MTP.
  Other Names: Bioelectrical impedance analysis

SUMMARY:
Background:

Dysphagia is frequently observed in subjects with chronic obstructive pulmonary disease (COPD). But tongue strength has not been investigated yet in COPD subjects. The investigators hypothesized that tongue strength is weaker in COPD subjects compared to normal subjects.

Methods:

This was a single-centre, observational, and cross-sectional study. Twenty-seven subjects with COPD and twenty-four age-matched control subjects were enrolled in this study. Isometric tongue strength was measured using a device fitted with a disposable oral balloon probe. The investigators also evaluated handgrip strength, gait speed, and appendicular skeletal muscle mass (ASM) to define participants as having sarcopenia. ASM, fat free mass index (FFMI), and skeletal muscle mass index (SMI) were measured by bioelectrical impedance analysis. Gait speed was measured using the 6-meter walking test. The eating assessment test-10 (EAT-10) was used to diagnose dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable COPD.
* Age-matched control subjects who did not have any pulmonary disease.

Exclusion Criteria:

* Participants with metallic implants.
* History of stroke disease.
* History of neuromuscular disease.
* Participants who did not have their front teeth.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: COPD subjects were chosen from a group of subjects who had visited the Department of Respiratory Medicine and Allergology at Kindai University Hospital from December 2019 to May 2020.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
maximum tongue pressure | 1 day
  To measure maximum tongue pressure (MTP), the balloon was positioned on the anterior palate with the lips closed. Subjects raised their tongue and compressed the balloon onto the palate with maximal voluntary muscular effort for approximately 7s. The measurement was taken three times with a 1-min interval. The maximum value was recorded as the MTP.

SECONDARY OUTCOMES:
handgrip strength | 1 day
  Handgrip strength was measured three times for the right hand using a grip strength dynamometer and mean values were used.
fat free mass index (FFMI) | 1 day
  FFMI (kg/m^2) was calculated by fat free mass／height^2(m^2).
skeletal muscle mass (SMI) | 1 day
  SMI (kg/m^2) was calculated by skeletal muscle mass ／height^2(m^2).
fat free mass | 1 day
  Fat free mass was measured using the medical body composition analyzer. It is designed for measurements in the supine position, using four pairs of electrodes (eight electrodes in total), positioned on each hand and foot21. Supine measurements were taken after lying down for 10 minutes. Alcohol was prohibited for 24h prior to the impedance measurements.
skeletal muscle mass | 1 day
  Skeletal muscle mass was measured using the medical body composition analyzer. It is designed for measurements in the supine position, using four pairs of electrodes (eight electrodes in total), positioned on each hand and foot21. Supine measurements were taken after lying down for 10 minutes. Alcohol was prohibited for 24h prior to the impedance measurements.
height | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Kindai University Faculty of Medicine, Ōsaka-sayama, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No